CLINICAL TRIAL: NCT02766140
Title: Multicentre, Randomised, Double-blind, Phase III Trial to Investigate the Efficacy and Safety of Oral SHR1020 Plus Docetaxel Therapy Compared to Placebo Plus Docetaxel Therapy in Patients With Local Advanced or Metastatic or Recurrent Non Squamous Non Small Cell Lung Cancer After Failure of First Line Chemotherapy.
Brief Title: SHR1020 Plus Docetaxel as Compared to Placebo Plus Docetaxel in 2nd Line Non Squamous Non Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: difficulty in recruitment
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-FMTN-II/III-NSCLC-COM
Record Dates: First submitted 2016-04-18; First posted 2016-05-09 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2018-12

CONDITIONS: Non Squamous Non Small Cell Lung
MeSH Terms: interventions — famitinib; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SHR1020 plus Docetaxel (Experimental)
  Interventions: Drug: SHR1020 plus Docetaxel
- Placebo plus Docetaxel (Placebo Comparator)
  Interventions: Drug: Placebo plus Docetaxel

INTERVENTIONS:
Drug: SHR1020 plus Docetaxel — SHR1020 20mg qd 2-21days, Docetaxel 60 mg/m^2 IV Day1/3weeks
  Arms: SHR1020 plus Docetaxel
Drug: Placebo plus Docetaxel — Placebo matching SHR1020 qd 2-21days, Docetaxel 60 mg/m^2 IV Day1/3weeks
  Arms: Placebo plus Docetaxel

SUMMARY:
The present trial will be performed to evaluate whether SHR1020 in combination with docetaxel in patients with Local Advanced or Metastatic or recurrent Non Squamous NSCLC is more effective as compared to placebo in combination with docetaxel. A secondary aim is to obtain safety information as well as information on quality of life of patients treated with SHR1020 in combination with docetaxel.

ELIGIBILITY:
Inclusion Criteria:

1. age:18-70 years
2. Histologically or cytologically confirmed locally advanced and/or metastatic NSCLC or recurrent NSCLC (≤9 months from date of diagnosis to randomized ), epidermal growth factor receptor-wild type, Anaplastic Lymphoma Kinase-wild type or unknown mutation
3. At least one lesion that can be accurately measured and has not been received local treatments such as radiotherapy and cryotherapy
4. Relapse or failure of one first line prior platinum-based chemotherapy
5. Eastern Cooperative Oncology Group performance status 0 or 1
6. Life expectancy of at least 12 weeks
7. Adequate organ and bone marrow function as defined below(no blood transfusion or drugs for leucopenia and Platelet within 14 days before screening): (1) HB≥90g/l (2) ANC≥1.5×10^9/l (3) PLT≥100×10^9/l (4) BIL<1.25×upper limit of normal (5) Alanine Aminotransferase and/or AST<2.5×upper limit of normal (< 5×upper limit of normal for patients with liver metastasis) (6) Cr≤1.25×upper limit of normal or Creatinine clearance rate>45ml/min ( Cockcroft-Gault Formula) (7) Cholesterol≤1.5×upper limit of normal, Triglyceride≤2.5×upper limit of normal (8) Left ventricular ejection fraction (LVEF) greater than lower limit of normal
8. Female: child bearing potential, a negative urine or serum pregnancy test result within 7 days before randomisation, agree to use effective contraception while on treatment and for at least 6 months after end of treatment;male: agree to use effective contraception while on treatment and for at least 6 months after end of treatment
9. Patient has given written informed consent

Exclusion Criteria:

1. More than one prior chemotherapy regimen for advanced and/or metastatic or recurrent NSCLC (except neoadjuvant or adjuvant chemotherapy )
2. Previous therapy with other VEGFR inhibitors、recombinant human endostatin、 docetaxel or immunotherapy for treatment of NSCLC
3. History of severe hypersensitivity reactions to docetaxel or other drugs formulated with polysorbate 80 (Tween 80), Hypersensitivity to the excipients of the trial drugs or contrast medium
4. Have clinically significant cavity effusion,such as pleural effusion、 pericardial effusion or ascites and require clinical intervention
5. Active brain metastases
6. Other malignancy within the past (including primary brain tumor or Leptomeningeal tumor), other than basal cell skin cancer or carcinoma in situ of the cervix
7. Significant weight loss (>10%) within the past 6 weeks
8. Persistence of clinically relevant therapy related toxicities from previous therapy (greater than Common Terminology Criteria for Adverse Event(CTCAE) 4.0 grade 1)
9. Treatment with surgery, chemotherapy, hormone therapy, radiotherapy, immunomodulation or monoclonal antibody therapy within the past 4 weeks and traditional chinese medicine for antitumor therapy within the past 2 weeks before start of therapy
10. Radiographical evidence of cavitary or necrotic tumours
11. Centrally located tumours with radiographical evidence (CT or MRI) of local invasion of major blood vessels
12. Greater than CTCAE 4.0 grade 2 pulmonary hemorrhage within the past one month before screening
13. History of clinically significant haemoptysis within the past 3 months (more than half a teaspoon within 24 hours )
14. History of major thrombotic or clinically relevant major bleeding event in the past 6 months
15. Prothrombin time (PT) and/or partial thromboplastin time (PTT) > 50% of devi

    * ation of upper limit of normal
16. Application of anticoagulants or vitamin K antagonists such as warfarin, heparin or its analogus, if INR≤1.5, with the purpose of prevention,the use of low-dose warfarin (1mg, qd) or aspirin ( ≤ 100 mg per day ) is allowed
17. Incomplete wound healing or fracture for long time
18. Uncontrolled hypertensin with one antihypertensive agent, unstable angina, history of myocardial infarction in the past 6 months, congestive heart failure>NYHA II, serious cardiac arrhythmia
19. Urinary protein≥++ and confirmed 24-hour urinary protein greater than 1.0g;
20. Preexisting thyroid dysfunction, even with medical therapy, thyroid function can not be maintained in the normal range
21. Uncontrolled diabetes mellitus with antidiabetic therapy
22. Current peripheral neuropathy greater than CTCAE 4.0 grade 2
23. Active or chronic hepatitis C and/or B infection with liver dysfunction
24. History of immunodeficiency diseases, other acquired or congenital immunodeficiency diseases, or history of organ transplantation
25. Serious infections requiring systemic antibiotic therapy
26. Variety of factors that affect the oral medication (such as unable to swallow, chronic diarrhea, bowel obstruction and other gastrointestinal disorders or abnormalities
27. Pregnancy or breast feeding
28. Active alcohol or drug abuse
29. Treatment in another clinical trial within the past 4 weeks before start of therapy
30. Psychological, familial, sociological, or geographical factors potentially hampering compliance with the study protocol and follow-up schedule
31. According to the investigator, other conditions that may increase the risk associated with patient safety and study participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Overall Survival | approximately 30 months

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | approximately 30 months
Incidence and Intensity of Adverse Events | From signing informed consent document until 30 days after the last drug administration
Objective Tumour Response (Complete Response Plus Partial Response) Using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | approximately 30months
Disease Control (Complete Response Plus Partial Response plus stable disease) Using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | approximately 30months
Quality of Life (QoL) measured by standardised questionnaires (EORTC Quality of Life Questionnaire-C30) | approximately 30months

CONTACTS AND LOCATIONS:
Overall Officials: caicun zhou, doctor, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China